CLINICAL TRIAL: NCT02716064
Title: Teams Advancing Patient Experience: Strengthening Quality for People With Cardiovascular and Metabolic Disease (TAPESTRY-CM): A Pilot Study
Brief Title: TAPESTRY for People With Cardiovascular and Metabolic Disease: A Pilot Study
Acronym: TAPESTRY-CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-450
Record Dates: First submitted 2014-12-03; First posted 2016-03-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: chronic conditions, self-management, PHR
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAP-CM Intervention (Experimental): Patients in this arm will be encouraged to complete the Healthy Lifestyle App modules and use McMaster PHR to self manage their chronic disease. Participants will also be completing the health and life goals using the App. The TAPESTRY-CM reports generated will then be reviewed by the clinic huddle teams
  Interventions: Behavioral: TAP-CM Intervention

INTERVENTIONS:
Behavioral: TAP-CM Intervention — The intervention includes: 1) Healthy Lifestyle App Goal Setting and Prioritization and modules, 2) TAP-CM Report triage Huddle with Interprofessional Team 3) The connection of patients to appropriate community resources 4) Volunteer helping with technology use

SUMMARY:
TAPESTRY-CM pilot study is a 12-week pilot test of the TAPESTRY-CM using a web application (APP) to help patient manage their diabetes and hypertension and other chronic conditions by assisting them in setting goals and connecting them to their healthcare team.

DETAILED DESCRIPTION:
This pilot study is a program evaluation that will employ developmental evaluation techniques to collect qualitative and quantitative data that will be handled, using a sequential explanatory mixed methods approach.Developmental evaluation is particularly useful for pre-formative development of potential scalable interventions. Developmental evaluation tracks and attempts to make sense of what emerges under conditions of complexity, documenting and interpreting the dynamics, interactions, and interdependencies that occur as innovations unfold. It will be helpful to explicitly understand: 1) what important decisions occur during the TAPESTRY-CM intervention development process and; 2) what data have validated those decisions about how the intervention will be structured and delivered. This understanding will provide a basis for describing key decisions and their rationale to our community and to other communities so that they make more informed adaptations to their local context.

TAPESTRY-CM has applied the principles of participatory design by engaging community stakeholders to co-create and refine TAPESTRY-CM interventions in the early phases of the project.

The use of mixed methods was purposefully chosen for this developmental evaluation. Answering a set of related research questions which included the collecting, analyzing and interpreting of qualitative and quantitative data increases the depth of understanding of results, provides stronger evidence for patterns or themes if data converge, can neutralize or cancel out some of the disadvantages of each method alone, and explicitly recognizes that social phenomena are complex such that varied methods are helpful to best understand these complexities.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 55 at the start of the study
* Patients with both diabetes and hypertension
* Patients with access to a computer and the internet

Exclusion Criteria:

* Patient is palliative or receiving end-of-life care
* Patient is deceased
* Has explicitly stated that they do not want to be part of a research project
* Patient resides in long-term care
* Patient has indicated that they do not want to receive a home visit from trained community volunteers.
* Patient or family member does not speak English
* Patient will be out of the country for more than 50% of trial duration
* Patients without access to a computer with the internet

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The experience of patients, family members, primary health care providers, volunteers and community organizations with the TAPESTRY-CM program | 12 weeks
  Qualitative measure and chart audit evaluating the experience of all participants in the pilot

SECONDARY OUTCOMES:
Experience of enrollment by patients | 12 weeks
  Qualitative measure - focus groups/interviews with patients
Extent volunteers needed to facilitate PHR set-up | 12 weeks
  Quantitaive measures: technology skills self-assessment scale (volunteers) scale, Qualitative measure: usability testing, and documentation of help-line inquiries
Burden on healthcare providers to respond to PHR queries from patients | 12 weeks
  Qualitative measure - focus groups and interviews with involved healthcare providers to assess the role of or burden on healthcare providers.
Patient interest in digital step tracking devise | 12 weeks
  Measure 1: yes/no data from App; Measure 2: qualitative- focus groups or interviews to test the usability of activity trackers.
Feasibility of using a structured goal setting process with patients including a formal Goal Attainment Scaling | 12 weeks
  Qualitative: focus groups or interviews and patient enablement scores; Quantitative: Using Goal Attainment Scales, to assess the usability of Goal Attainment Scaling;
Developmental decision evaluation - I | 12 weeks
  mportant decisions during the TAPESTRY-CM intervention development process that affected initial implementation or changes in delivery of the TAP-CM intervention and what data supported the decisions made. Using a template to record the number and type of decisions, assessed using qualitative and quantitative analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Family Practice, Hamilton, Ontario
  - Stonechurch Family Health Centre (SFHC), Hamilton, Ontario